CLINICAL TRIAL: NCT06715709
Title: Corticosteroids in Total Knee Arthroplasty: How Many Dexamethasone Doses Should Be Given Perioperatively? A Randomized Controlled Trial
Brief Title: How Many Dexamethasone Doses Should Be Given Perioperatively?
Acronym: DEXA_PERIOP
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Charles P. Hannon, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 24-008239
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Arthropathy of Knee

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- (1) dexamethasone administered intraoperatively at the time of anesthesia (Other): (1) dexamethasone administered intraoperatively at the time of anesthesia
  Interventions: Drug: Dexamethasone IV
- (2) dexamethasone administered intraoperatively and on the morning of the first postoperative day, (Experimental): (2) dexamethasone administered intraoperatively and on the morning of the first postoperative day,
  Interventions: Drug: Dexamethasone IV+Oral
- (3) dexamethasone administered intraoperatively, the morning of the first& second postoperative day (Experimental): (3) dexamethasone administered intraoperatively, the morning of the first postoperative day, and the morning of the second postoperative day.
  Interventions: Drug: Dexamethasone IV+Oral 2 Day

INTERVENTIONS:
Drug: Dexamethasone IV — Patients will receive dexamethasone administered intraoperatively at the time of anesthesia. The dose of dexamethasone will be 16mg intravenous (IV) if you do not have a prior diagnosis of diabetes mellitus, or 8mg IV if you do have a previous diagnosis of diabetes mellitus.
  Arms: (1) dexamethasone administered intraoperatively at the time of anesthesia
Drug: Dexamethasone IV+Oral — Patients will receive dexamethasone administered intraoperatively and on the morning of the first postoperative day. The dose of dexamethasone will be 16mg intravenous (IV) if you do not have a prior diagnosis of diabetes mellitus, or 8mg IV if you do have a previous diagnosis of diabetes mellitus. The medication will be intravenously administered while inpatient, and via oral route when discharged.
  Arms: (2) dexamethasone administered intraoperatively and on the morning of the first postoperative day,
Drug: Dexamethasone IV+Oral 2 Day — Patients will receive dexamethasone administered intraoperatively, the morning of the first postoperative day, and the morning of the second postoperative day. The dose of dexamethasone will be 16mg intravenous (IV) if you do not have a prior diagnosis of diabetes mellitus, or 8mg IV if you do have a previous diagnosis of diabetes mellitus. The medication will be intravenously administered while inpatient, and via oral route when discharged.
  Arms: (3) dexamethasone administered intraoperatively, the morning of the first& second postoperative day

SUMMARY:
The purpose of this study is to determine the most efficient and safest dexamethasone dose given perioperatively during total knee arthroplasty that reduces postoperative option consumption and pain, improves postoperative nausea and vomiting, and minimizes postoperative complications

DETAILED DESCRIPTION:
Perioperative multimodal analgesia and anesthesia regimens have become the standard of care in modern total joint arthroplasty. This has been driven in part by an emphasis on decreasing postoperative opiate use, a growing trend towards shorter inpatient hospital stays and outpatient TKAs, and motivation to improve patient satisfaction after TKA. Acute postoperative pain not only decreases patient satisfaction,1 but can also lead to associated complications including chronic opioid use,2 disrupted sleep,3 and impaired early mobilization, which can prolong recovery and increase the risk of medical complications such as venous thromboembolism (VTE).4,5 Previously, opioids were the basis of pain management regimens, however, opioids may cause significant adverse events including nausea, vomiting, ileus, sedation, urinary retention, respiratory depression, and others, in addition to a risk of addiction.6 Conversely, contemporary arthroplasty relies on minimizing opiate use by administering multimodal analgesia and anesthesia that target various pain and inflammatory pathways7,8 to improve postoperative outcomes and facilitate rapid discharge postoperatively.

Corticosteroids are potent anti-inflammatory medications with anti-emetic properties,9,10 with previous studies demonstrating their effectiveness in reducing postoperative pain, nausea, and vomiting.9 Therefore, corticosteroids are commonly used in current multimodal pain management regimens. Dexamethasone is one of the most well-studied corticosteroids in the total joint arthroplasty literature. Previous randomized controlled trials evaluated the administration of multiple perioperative dexamethasone doses compared to one dose of perioperative dexamethasone and reported that multiple doses were associated with reduced opioid consumption and pain in the early postoperative period after TKA,11-13 while another reported no significant differences.14 Furthermore, while Xu et al. did not demonstrate a difference in postoperative nausea and vomiting between patients receiving one perioperative dexamethasone dose versus three doses,13 other RCTs reported that additional doses of dexamethasone was associated with significantly decreased postoperative nausea.11,12 This is important because postoperative nausea is a commonly cited adverse effect of anesthesia. The RCT by Xu et al. compared one dose to three doses of dexamethasone,13 while the RCTs by Backes et al., Wu et al., and Gasbjerg et al. compared one dose to two doses of dexamethasone in the setting of TKA.11,12,14 Following total hip arthroplasty, Lei et al. evaluated two doses of perioperative dexamethasone to three doses and reported that the three dose treatment arm had greater reductions in postoperative pain and nausea, greater range of motion, and shorter length of hospital stays, without any increase in adverse events.15 To our knowledge, there is no randomized controlled trial directly comparing multiple-dose treatment arms (i.e. one versus two versus three or more perioperative dexamethasone doses) in the setting of TKA. Therefore, the standard number of doses of dexamethasone that should be administered in the perioperative period has not been established.

Furthermore, concern remains regarding the theoretical adverse events that may be associated with corticosteroid administration, including decreased wound healing, increased risk of infection, or gastrointestinal hemorrhage.16,17 Previous studies investigating dexamethasone may have excluded patients with diabetes mellitus or poorly controlled diabetes mellitus due to concern that corticosteroids would increase blood glucose levels, thereby increasing the risk of medical complications or periprosthetic joint infection. However, while some studies have demonstrated corticosteroid use may lead to transient increases in blood glucose levels, recent studies have reported no difference in postoperative complication rates.13,18,19 Heterogeneity between studies, small sample sizes, and exclusion of at-risk groups, such as diabetic patients, limit many previous studies that reported on complications associated with corticosteroid use in total joint arthroplasty. Further research is required to characterize the safety profile of dexamethasone in patients receiving TKA.

The previous literature is heterogenous in the dose, number of doses, and timing of perioperative dexamethasone that was administered, in addition to a lack of standardization in the multimodal analgesia and anesthesia regimen. Therefore, the purpose of this study is to perform a multicenter randomized controlled trial to determine the optimal number of dexamethasone doses to be administered in the TKA perioperative period by comparing postoperative outcomes in patients receiving one, two, or three doses of intravenous dexamethasone.

ELIGIBILITY:
Inclusion Criteria

* Age > 18 years
* Primary total knee arthroplasty

Exclusion Criteria

* Age < 18 year
* Revision or unicompartmental knee arthroplasty
* Corticosteroid use within 3 months prior to TKA
* Inflammatory arthritis
* Current systemic fungal infection
* Renal or liver failure
* Prior adverse reaction to corticosteroid
* Primary TKA requiring hardware removal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | 72 hours
  Cumulative opioid consumption within 72 hours after Total Knee Arthroplasty, measured in oral morphine milligram equivalents.

SECONDARY OUTCOMES:
Sleeplesssness | 7 days
  Sleeplessness will be measured by recording the number of hours slept in a 24-hour period for 7 days postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Hannon, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No